CLINICAL TRIAL: NCT01818674
Title: Microclinic Social Network Behavioral Health Trial for Obesity and Metabolic Risk Factor Control in Jordan
Brief Title: Microclinic Social Network Behavioral Health Trial in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microclinic International (Other)
Collaborators: Royal Health Awareness Society (RHAS) (Unknown); Jordanian Ministry of Health (MoH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WDF2010-2014
Record Dates: First submitted 2013-03-05; First posted 2013-03-26 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Hypertension; Hyperglycemia; Blood Pressure; Hyperglycaemia (Diabetic); Body Weight; Weight Loss; Weight, Body; Weight Change Trajectory; Weight Change, Body; Weight Gain; Blood Pressure, High; Social Behavior; Behavior, Health; Lifestyle Risk Reduction; Lifestyle, Healthy; Diabetes; Diabetes Mellitus; Glucose, High Blood
Keywords: social network; microclinic; middle east; jordan; intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertension; Hyperglycemia; Body Weight; Weight Loss; Body-Weight Trajectory; Body Weight Changes; Weight Gain; Social Behavior; Health Behavior; Risk Reduction Behavior; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Microclinic Behavioral Health Enhanced Program (Experimental): Group A received the Microclinic Behavioral Health Full Program (structured social interactions + fully interactive classroom education curriculum; parallel clinical screenings)
  Interventions: Behavioral: Microclinic Behavioral Health Full Program (education curriculum in classroom setting, plus full social interaction program)
- Group B - Microclinic Behavioral Health Basic Program (Experimental): Group B received the Microclinic Behavioral Health Basic Program (no social structured interactions; basic classroom education; parallel clinical screenings)
  Interventions: Behavioral: Microclinic Behavioral Health Basic Program (education-only in classroom setting; no structured social interactions)
- Group C - Controls with Parallel Monitoring (No Intervention): Group C only received standard care, and only received parallel risk factor screening measurements; not participation in classroom or any social activities.

INTERVENTIONS:
Behavioral: Microclinic Behavioral Health Full Program (education curriculum in classroom setting, plus full social interaction program) — A 6-month intervention program (sessions and educational materials) aims to increase knowledge and skills in diabetes self-management and peer support and monitoring. The curriculum include causes of diabetes, prevention of complications, symptoms, self-management strategies, diet, exercise, peer monitoring and support by trained Project nurses from MoH health centers, local physicians, and university professors. Each class will provide 2-3 hours of discussion to foster active class participation and engagement.
  Other Names: Group A
  Arms: Group A - Microclinic Behavioral Health Enhanced Program
Behavioral: Microclinic Behavioral Health Basic Program (education-only in classroom setting; no structured social interactions) — This basic program (6 month) aims to increase participants knowledge about diabetes self-management, but without structured social interaction programming. While group classroom setting is still used for delivery of the educational curriculum, the education program in group B have no group-based or team-building activities, group goal setting, and classroom program is lecture style with more limited class participation and interaction.
  Other Names: Group B
  Arms: Group B - Microclinic Behavioral Health Basic Program

SUMMARY:
This 3-armed randomized controlled trial aims to evaluate the effectiveness of The Microclinic Behavioral Health Program in improving obesity and diabetes risk factors through a behavioral intervention program structured to enhance and promote social-network interactions and social support. The full version of the Microclinic Behavioral Health Program (Full MCP) with program-activated social-network interactions-with shared access to diabetes education, technology, and group support to promote weight and metabolic control through diet, exercise, medication adherence, and blood pressure management. Participants play a role in the collective effort to combat diabetes and solidifying self-management behavioral skills through peer-monitoring and encouragement of lifestyle behaviors. The study may yield valuable information on the impact of social support and social network interactions for enhancing body weight and blood sugar control. We compare the full MCP intervention, to a basic MCP intervention with more limited classroom interaction, and to an parallel monitoring control arm. And we aim to understand how metabolic changes over time relate to the cross-propagation of health behaviors between persons in social networks.

This Microclinic Behavioral Health Program was established in collaboration with the Royal Health Awareness Society (RHAS) and the Jordanian Ministry of Health (MoH).

DETAILED DESCRIPTION:
I. Objectives

Because social network-based programs have shown promise as a viable public health intervention strategy, we designed the MCP program to leverage existing social relationships to propagate positive health behaviors in efforts to prevent and manage obesity and diabetes. We conduct a trial to examine the effectiveness of the Microclinic Behavioral Health Program via 3 arm trial in Jordan of a 6 month intervention with 2 years followup.

Furthermore, we aim to uncover the social mechanism of the intervention -- notably to define the pathways through which the social network behavioral health program worked by partitioning the different social network processes of direct causal induction (i.e. change catalyzed by a social network) from homophilly (i.e. where social networks are formed based on similar health behaviors), and confounding (i.e. correlation with exogenous shared variable). Notably, we seek to determine the presence of the amplification of metabolic changes over time due to the cross-propagation of health behaviors between persons in a social network.

II. Study Design

Randomized Control Study: This study is a randomized control study of adults (>= 18 years old) with Type 2 diabetes mellitus, pre-diabetes, or at risk for diabetes, who will be randomly assigned to an intervention group consisting of the Microclinic Behavioral Health Enhanced Program (Group A), a group who will receive the Microclinic Behavioral Health Basic Program without the social network components (Group B) , and controls receiving standard care and risk factor monitoring (Group C).

III. Study Procedures

a. Participant Recruitment (1-3 months) The aim of recruitment is to inform individuals with diabetic, pre-diabetic, or at risk for diabetes in the community about the microclinic study, and encourage patients to participate. The recruitment process will consist of interconnected strategies including: 1) the distribution of posters and invitations in four catchment areas, and a broader media campaign, and 2) recruitment by nurses through clinics in two pilot locations around Amman.

Recruitment: Outreach strategies to recruit patients at risk for diabetes and with Type 2 diabetes include: a) The Royal Health Awareness Society will lead an outreach effort to spread the word about the Microclinic Social Network Behavioral Health Trial. The effort will involve distribution of posters and flyers in the public sphere, and, if possible, airing of radio or television spots. b) At the three assigned Ministry of Health local health centers, a Project Officer for each center will work with Project nurses trained in research, Institutional Review Board approved protocol, and data collection to recruit patients at risk for diabetes, pre-diabetes, and with type 2 diabetes to the Microclinic Social Network Behavioral Health Trial.

Potential participants, consisting of both local residents and refugees in Jordan will be contacted by phone or referred to the trial in person during their visit to local Jordan Ministry of Health centers and asked if they would be willing to participate.

Group A shall receive the 6 month Microclinic Behavioral Health Full Program, via trained Project Nurses, and a classroom curriculum that will increase the knowledge and skills in diabetes self-management and peer support and monitoring. The educational curriculum includes sessions on the causes of diabetes, prevention of complications, symptoms, self-management strategies, diet, exercise, but with emphasis on peer monitoring, social support, and structured social interactions. Each session is 2-3 hours.

Group B receiving a modified Microclinic Behavioral Health Basic Program that has the same educational curriculum and classroom setting, but a modified version that does not emphasize the importance of social support, without structured social interaction enhancing components. Group C receiving no intervention and therefore, standard care as the control group, with parallel measurement of risk factors (to alleviate monitoring bias).

A critical component of this project is the evaluation aimed at assessing the long term efficacy and sustainability of the Microclinic interventions in improving body weight and glucose in a resource limited setting over a 2 year time span. The program evaluation will collect demographic, medical history, clinical data, behavioral data from all participants during the 6 month main program as well as at 2 years after baseline.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with type 2 diabetes, pre-diabetes, or 'at-risk for diabetes' (defined below)
2. live in the catchment area of the study
3. provide informed consent to participate.

Exclusion Criteria:

1. participants who are not diagnosed with type 2 diabetes, pre-diabetes, or 'at-risk for diabetes'
2. are not able to provide informed consent due to mental illness
3. women who are pregnant.

   * Pregnant women may participate in consultation with their physician. However, data related to their participation in the trial will not be included in data analysis.

'At-risk of diabetes' is defined as either: a) having a history of diabetes in close family AND being overweight/obese, or b) having a family history of diabetes AND having either high BP or high serum cholesterol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in body weight across all trial arms, over entire study | Overall change across baseline, to 6 months, to 2 years
  Change in body weight from baseline, a joint test of differences across all trial arms
Longitudinal change in fasting blood glucose across all trial arms, over entire study | Overall change across baseline, to 6 months, to 2 years
  Change in fasting blood glucose from baseline, a joint test of differences across all trial arms
Longitudinal change in glycosylated hemoglobin (HbA1c) across all trial arms, over entire study | Overall change across baseline, to 6 months, to 2 years
  Change in HbA1c from baseline, a joint test of differences across all trial arms
Longitudinal change in blood pressure across all trial arms, over entire study | Overall change across baseline, to 6 months, to 2 years
  Change in mean arterial pressure (indexed from systolic and diastolic blood pressure) from baseline, a joint test of differences across all trial arms. mean arterial pressure was calculated using the clinical formula MAP=(SBP + (2*DBP))/3)
Temporally investigate the causal induction of cascading changes in body weight between follow-ups on subsequent weight changes in other participants. | Change from each session (weekly, biweekly, triweekly), on each subsequent session, during 6 month intervention period.
  Using time intervals between follow-ups analyzed as separate induction timeframe windows, we estimate how weight loss observed in a previous time window predicts body weight change in subsequent followup intervals of the other participants.

SECONDARY OUTCOMES:
Relative changes in body weight between individual trial arms | Change from baseline, at 6 months, at 2 years
  Cross comparisons in longitudinal change in body weight between A vs. C, B vs. C, A vs. B.
Relative changes in fasting glucose between individual trial arms | Change from baseline, at 6 months, at 2 years
  Cross comparisons in longitudinal change in fasting glucose between A vs. C, B vs. C, A vs. B.
Relative changes in HbA1c between individual trial arms | Change from baseline, at 6 months, at 2 years
  Cross comparisons in longitudinal change in HbA1c between A vs. C, B vs. C, A vs. B.
Relative changes in blood pressure between individual trial arms | Change from baseline, at 6 months, at 2 years
  Cross comparisons in longitudinal change in mean arterial pressure (indexed from systolic and diastolic blood pressure) between A vs. C, B vs. C, A vs. B. (mean arterial pressure was calculated using the clinical formula MAP=(SBP + (2*DBP))/3)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Zoughbie, D.Phil., Principal Investigator — Microclinic International; Eric L Ding, Sc.D., Principal Investigator — New England Complex Systems Institute
Locations (3):
- Jordan (3):
  - Abu Nseir Ministry of Health Center, Amman
  - Kreibet Al Souq Ministry of Health Center, Amman
  - Naour Ministry of Health Center, Amman

REFERENCES:
- [Derived] Ding EL, Feigl AB, Watson KT, Ng TLJ, Makerechi L, Bui N, Ireifij A, Farraj R, Zoughbie DE. Social network enhanced behavioral interventions for diabetes and obesity: A 3 arm randomized trial with 2 years follow-up in Jordan. PLOS Glob Public Health. 2024 Mar 20;4(3):e0001514. doi: 10.1371/journal.pgph.0001514. eCollection 2024. PMID 38507441
- See also: Microclinic International homepage — http://microclinics.org